CLINICAL TRIAL: NCT07310472
Title: Administration of the Nasal Influenza Vaccine to Children in Daycare or at a Healthcare Facility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: T2025/11144
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Influenza Vaccination
Keywords: Influenza; Children; Vaccination coverage; Nasal influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Cluster-randomized study, daycare units being clusters for randomization. Data collection from the vaccination registry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants are offered a nasal influenza vaccine at daycare
  Interventions: Behavioral: Possibility to get live attenuated nasal influenza vaccine at daycare
- Comparison group (No Intervention): Participants are not offered a nasal influenza vaccine at daycare

INTERVENTIONS:
Behavioral: Possibility to get live attenuated nasal influenza vaccine at daycare — The intervention is the possibility to get influenza vaccine in the daycare, in comparison to routine practice of getting influenza vaccine in a healthcare setting.
  Arms: Intervention group

SUMMARY:
The goal of this intervention study is to learn if giving children influenza vaccinations in early childhood education facilities (i.e., daycare) will increase vaccination coverage compared to giving vaccinations only at healthcare. The main question it aims to answer is:

• Does offering children nasal influenza vaccine in daycare result in higher proportion of children getting influenza vaccine.

Researchers will compare daycare setting and healthcare setting as the location of giving influenza vaccines to children to see if more children will get vaccinated if they have an opportunity to receive nasal influenza vaccine at daycare.

Participants in the intervention group will:

• Have the opportunity to receive influenza vaccine in the daycare or in the healthcare

Participants in the comparison group will:

• Have the opportunity to receive influenza vaccine in the healthcare only

ELIGIBILITY:
Inclusion Criteria:

* Attending early childhood education (daycare) in the city of Turku

Exclusion Criteria:

* No exclusion criteria

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6000 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Influenza vaccination coverage | From enrollment to the end of seasonal influenza vaccinations about 3 to 10 weeks later.
  Study child receiving any influenza vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No
According to national regulations, it is not allowed to share individual health data.